CLINICAL TRIAL: NCT03554278
Title: Alteration of Stool Microbiota in Preterm Infants Less Than 32 Weeks With Anemia, and Following Blood Transfusion
Brief Title: Alteration of Stool Microbiota in Preterm Infants With Anemia
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Julie Mirpuri Hathiramani, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 092017-028
Record Dates: First submitted 2018-05-03; First posted 2018-06-13 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Anemia, Neonatal; Necrotizing Enterocolitis; Dysbiosis
Keywords: NEC; transfusion; microbiome; premature
MeSH Terms: conditions — Anemia, Neonatal; Enterocolitis, Necrotizing; Dysbiosis; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anemia: Stool samples from infants with anemia. Severe anemia defined as hematocrit less than 25%. Anemia defined as hematocrit greater than or equal to 25% and less than 30%.
- No Anemia: Stool samples from infants without anemia. No anemia defined as hematocrit equal to or greater than 30%.

SUMMARY:
This study evaluates the relationship between anemia and stool microbiota in premature infants. It also evaluates the relationship between blood transfusion and stool microbiota.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is a leading cause of death in preterm infants, yet the disease mechanism is not well understood. Among the factors that have been studied are the change in stool microbiota (dysbiosis), severe anemia, and transfusion. Studies suggest that dysbiosis occurs in neonates with NEC. Large studies and meta-analyses have shown a predominance of Gammaproteobacteria, a decrease in Firmicutes, and decreased bacterial diversity in stool from infants with NEC. Studies do not support a relationship between transfusions and NEC since there are conflicting findings on this topic. There is a suggestion, however, that severe anemia may be associated with NEC though this requires further study.

No studies have been done evaluating the relationship between anemia and change in stool microbiota, or blood transfusion and change in stool microbiota. This study aims to primarily evaluate the relationship between anemia and stool microbiota, and secondarily evaluate the relationship between transfusion and stool microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 32 weeks gestation at birth
* Age at enrollment between 7 days and less than/equal to 30 days
* Minimum 100 mL/kg/day enteral feeds

Exclusion Criteria:

* Development of necrotizing enterocolitis (NEC) prior to enrollment
* Prior surgery
* Major congenital anomalies
* Oxygen requirement with FiO2 (fraction of inspired oxygen) >50% (at time of enrollment)

Ages: 7 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will enroll preterm infants that are less than 32 weeks gestational age at birth. At time of enrollment, these infants must be between 7 days of age up to (and including) 30 days of age. They must also be on enteral feeds of at least 100mL/kg/day. The investigators will exclude infants who have developed NEC prior to enrollment, who have had surgery prior to enrollment, who have major congenital anomalies, or who are requiring FiO2 >50% at time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
qRT-PCR (polymerase chain reaction) quantitative stool analysis | qRT-PCR will be analyzed for infant stool samples from enrollment until infants are 38 weeks corrected, or until they are discharged from the hospital. This time frame will be an average of 10 weeks per infant.
  Quantify major bacterial groups, including Proteobacteria, Firmicutes, and Bacteroides in stool samples

SECONDARY OUTCOMES:
Alpha diversity | Infant stool samples will be analyzed from enrollment until infants are 38 weeks corrected, or until they are discharged from the hospital. This time frame will be an average of 10 weeks per infant.
  Use next generation sequencing to assess changes in alpha diversity of bacteria between non-anemic and anemic stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Julie Mirpuri Hathiramani, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gritz EC, Bhandari V. The human neonatal gut microbiome: a brief review. Front Pediatr. 2015 Mar 5;3:17. doi: 10.3389/fped.2015.00017. eCollection 2015. PMID 25798435
- [Background] Patel RM, Denning PW. Intestinal microbiota and its relationship with necrotizing enterocolitis. Pediatr Res. 2015 Sep;78(3):232-8. doi: 10.1038/pr.2015.97. Epub 2015 May 20. PMID 25992911
- [Background] Warner BB, Tarr PI. Necrotizing enterocolitis and preterm infant gut bacteria. Semin Fetal Neonatal Med. 2016 Dec;21(6):394-399. doi: 10.1016/j.siny.2016.06.001. Epub 2016 Jun 22. PMID 27343151
- [Background] Warner BB, Deych E, Zhou Y, Hall-Moore C, Weinstock GM, Sodergren E, Shaikh N, Hoffmann JA, Linneman LA, Hamvas A, Khanna G, Rouggly-Nickless LC, Ndao IM, Shands BA, Escobedo M, Sullivan JE, Radmacher PG, Shannon WD, Tarr PI. Gut bacteria dysbiosis and necrotising enterocolitis in very low birthweight infants: a prospective case-control study. Lancet. 2016 May 7;387(10031):1928-36. doi: 10.1016/S0140-6736(16)00081-7. Epub 2016 Mar 9. PMID 26969089
- [Background] Zhou Y, Shan G, Sodergren E, Weinstock G, Walker WA, Gregory KE. Longitudinal analysis of the premature infant intestinal microbiome prior to necrotizing enterocolitis: a case-control study. PLoS One. 2015 Mar 5;10(3):e0118632. doi: 10.1371/journal.pone.0118632. eCollection 2015. PMID 25741698
- [Background] Pammi M, Cope J, Tarr PI, Warner BB, Morrow AL, Mai V, Gregory KE, Kroll JS, McMurtry V, Ferris MJ, Engstrand L, Lilja HE, Hollister EB, Versalovic J, Neu J. Intestinal dysbiosis in preterm infants preceding necrotizing enterocolitis: a systematic review and meta-analysis. Microbiome. 2017 Mar 9;5(1):31. doi: 10.1186/s40168-017-0248-8. PMID 28274256
- [Background] Patel RM, Knezevic A, Shenvi N, Hinkes M, Keene S, Roback JD, Easley KA, Josephson CD. Association of Red Blood Cell Transfusion, Anemia, and Necrotizing Enterocolitis in Very Low-Birth-Weight Infants. JAMA. 2016 Mar 1;315(9):889-97. doi: 10.1001/jama.2016.1204. PMID 26934258
- [Background] Hay S, Zupancic JA, Flannery DD, Kirpalani H, Dukhovny D. Should we believe in transfusion-associated enterocolitis? Applying a GRADE to the literature. Semin Perinatol. 2017 Feb;41(1):80-91. doi: 10.1053/j.semperi.2016.09.021. Epub 2016 Nov 17. PMID 27866662

DOCUMENTS (1):
  • Study Protocol (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03554278/Prot_000.pdf